CLINICAL TRIAL: NCT05945173
Title: Clinical Evaluation of the Effect of the Prolonged Evaporation Time of the Solvent of Two Universal Adhesives in Restorations of Non-carious Cervical Lesions: Double-blind Randomized Clinical Trial
Brief Title: Evaluation of the Solvent Evaporation Time of Universal Adhesives in the Quality of Cervical Lesions Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Principal Investigator, Mario Felipe Gutiérrez Reyes, Associate Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEC2022129
Record Dates: First submitted 2023-06-12; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Non-carious Cervical Lesions
Keywords: Dental bonding; Tooth erosion; Tooth wear; Adhesive systems; Solvent
MeSH Terms: conditions — Tooth Erosion; Tooth Wear

STUDY DESIGN:
Intervention Model Description: This is a four-arm, double-blind, randomized controlled clinical trial. Experimental group 1: 35 non-carious cervical lesions (NCCL) using an alcohol- and water-based solvent universal adhesive with evaporation of solvent for 25 seconds. Experimental group 2: 35 NCCL using an acetone-based universal solvent adhesive with solvent evaporation for 25 seconds. Control group 1: 35 NCCL using an alcohol- and water-based universal solvent adhesive with evaporation of solvent for 5 seconds. Control group 2: 35 NCCL using an acetone-based universal solvent adhesive with solvent evaporation for 5 seconds. LCNCs will be randomized to universal adhesive usage and evaporation time.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Two blinded, experienced, and calibrated dentists (who specialized in esthetic dentistry with more than 15 years of clinical practice), will perform the clinical evaluation. Patients will be also blinded to group assignment. An inter-examiner and inter-examiner agreement of at least 85% will be necessary before beginning the evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group 1 (Experimental): 35 non-carious cervical lesions (NCCL) will receive composite resin restorations in the selective enamel etching strategy.
  Interventions: Procedure: Evaporation time for 25 seconds; Device: alcohol/water-based universal adhesive
- Experimental group 2 (Experimental): 35 non-carious cervical lesions (NCCL) will receive composite resin restorations in the selective enamel etching strategy.
  Interventions: Procedure: Evaporation time for 25 seconds; Device: acetone-based universal adhesive
- Control group 1 (Active Comparator): 35 non-carious cervical lesions (NCCL) will receive composite resin restorations in the selective enamel etching strategy.
  Interventions: Procedure: Evaporation time for 5 seconds; Device: alcohol/water-based universal adhesive
- Control group 2 (Active Comparator): 35 non-carious cervical lesions (NCCL) will receive composite resin restorations in the selective enamel etching strategy.
  Interventions: Procedure: Evaporation time for 5 seconds; Device: acetone-based universal adhesive

INTERVENTIONS:
Procedure: Evaporation time for 5 seconds — Composite resin restorations of non-carious cervical lesions will be performed with an adhesive with solvent evaporation for 5 seconds.
  Other Names: Evaporation time of solvent for 5 seconds
  Arms: Control group 1; Control group 2
Procedure: Evaporation time for 25 seconds — Composite resin restorations of non-carious cervical lesions will be performed with an adhesive with solvent evaporation for 25 seconds.
  Other Names: Evaporation time of solvent for 25 seconds
  Arms: Experimental group 1; Experimental group 2
Device: alcohol/water-based universal adhesive — Composite resin restorations of non-carious cervical lesions will be performed with an alcohol/water-based universal adhesive (Scotchbond Universal Plus; 3M).
  Other Names: alcohol/water-based adhesive
  Arms: Control group 1; Experimental group 1
Device: acetone-based universal adhesive — Composite resin restorations of non-carious cervical lesions will be performed with an acetone-based universal adhesive (Gluma Universal Bond; Kulzer).
  Other Names: acetone universal adhesive
  Arms: Control group 2; Experimental group 2

SUMMARY:
The aim of this study will be to evaluate the effect of prolonging solvent evaporation time on the 6- and 12-months clinical performance of two universal adhesive systems used as selective enamel etch (SEE).

Methods: 140 restorations will be randomly placed in 35 subjects according to the following groups: SUP5 (Scotchbond Universal Plus evaporated for 5 s); SUP25 (Scotchbond Universal Plus evaporated for 25 s); GBU5 (Gluma Bond Universal evaporated for 5 s); GBU25 (Gluma Bond Universal evaporated for 25 s). Resin composite will be placed incrementally and light-cured. The restorations will be evaluated at baseline, after a week, 6 and 12 months using the FDI and USPHS criteria. Statistical analyses will be performed using appropriate tests (α = 0.05).

DETAILED DESCRIPTION:
This is a four-arm, double-blind, randomized controlled clinical trial. Experimental group 1: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations using an alcohol- and water-based solvent universal adhesive (Scotchbond Universal Plus; 3M) in the selective enamel etching strategy with evaporation of solvent for 25 seconds. Experimental group 2: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations using an acetone-based universal solvent adhesive (Gluma Universal Bond; Kulzer) in the selective enamel etching strategy with solvent evaporation for 25 seconds. Control group 1: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations, using an alcohol- and water-based universal solvent adhesive (Scotchbond Universal Plus; 3M), in the selective enamel etching strategy, with evaporation of solvent for 5 seconds. Control group 2: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations, using an acetone-based universal solvent adhesive (Gluma Universal Bond; Kulzer), in the strategy of selective enamel etching, with solvent evaporation for 5 seconds. LCNCs will be randomized to universal adhesive usage and flash-off time. All groups will be light-cured with a light-curing device (SmartLite Focus, Dentsply) with a light intensity of 855 mW/cm² for 20 seconds. Operators will restore the cervical area by applying three increments of resin (Opallis, FGM Prod. Odont.Ltda, Joinville, SC, Brazil). Each increment will light cure for 10 s at 1200 mW/cm2 (Radii Cal, SDI, Victoria, Australia). Restorations will be finished immediately with fine diamond burs (#3195F and #3195FF, KG Sorensen, Barueri, SP, Brazil) and polished with discs and polishing gums (Soflex, 3 M ESPE, St. Paul, MN, EE. UU.).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Presence of at least two Non-Carious Cervical Lesions in the dental arch with a need for restorative treatment.
* Acceptable level of oral hygiene according to the Simplified Oral Hygiene Index.
* At least 20 teeth in function.
* Non-Carious Cervical Lesions with a maximum of 50% of enamel margin.

Exclusion Criteria:

* Driving difficulties that prevent adequate oral hygiene.
* Periodontal disease.
* Active caries lesions on the teeth included in the research.
* Parafunctional habits.
* Active staples of removable partial dentures on the teeth included in the research and that these are not pillars of prostheses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Retention of restorations | From date of randomization until twenty four months
  Retention measured by World Dental Federation (FDI) criteria as following:
  * VG: Clinically very good - Restoration retained, no fractures / cracks;
  * G: Clinically good - Small hairline crack;
  * SS: Clinically sufficient/satisfactory - Two or more or larger hairline cracks and/or chipping (not affecting the marginal integrity);
  * US: Clinically unsatisfactory - Chipping fractures which damage marginal quality; bulk fractures with or without partial loss (less than half of the restoration);
  * PO: Clinically poor - (Partial or complete) loss of restoration, (replacement necessary).

SECONDARY OUTCOMES:
Marginal Adaptation of restorations | From date of randomization until twenty four months
  Marginal Adaptation measured by World Dental Federation (FDI) criteria as following:
  * VG: Clinically very good - Harmonious outline, no gaps, no discoloration;
  * G: Clinically good - Small marginal fracture removable by polishing;
  * SS: Clinically sufficient/satisfactory - Several small enamel or dentin fractures;
  * US: Clinically unsatisfactory - Notable enamel or dentine wall fracture;
  * PO: Clinically poor - Filling is loose but in situ.
Marginal Staining of restorations | From date of randomization until twenty four months
  Marginal Staining measured by World Dental Federation (FDI) criteria as following:
  * VG: Clinically very good - No marginal staining;
  * G: Clinically good - Minor marginal staining, easily removable by polishing;
  * SS: Clinically sufficient/satisfactory - Moderate marginal staining, not esthetically unacceptable;
  * US: Clinically unsatisfactory - Pronounced marginal staining; major intervention necessary for improvement;
  * PO: Clinically poor - Deep marginal staining not accessible for intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mario Felipe Gutiérrez Reyes, PhD, Study Director — Universidad de los Andes, Chile
Locations (1):
- Mario Felipe Gutiérrez Reyes, Santiago, Santiago Metropolitan, Chile